CLINICAL TRIAL: NCT04372914
Title: Effect of Oral Black Raspberry Administration on Oral Cell DNA Adducts in Smokers
Brief Title: Prevention of Oral DNA Damage by Black Raspberries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karam El-Bayoumy, Associate Director for Basic Research, Penn State Cancer Institute, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00013621; R01CA173465 (NIH)
Record Dates: First submitted 2020-04-22; First posted 2020-05-04 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Oral Cancer; Smoking; DNA Damage; Oxidative Stress
MeSH Terms: conditions — Mouth Neoplasms; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRB Lozenges (Experimental): Oral lozenges that contain 1 gram of BRB freeze-dried powder
  Interventions: Dietary Supplement: BRB Lozenges

INTERVENTIONS:
Dietary Supplement: BRB Lozenges — Each lozenge is made from 1 gram of freeze-dried black raspberry powder (equivalent to ~5 black raspberries) in the form of a dissolvable slow-release lozenge.

SUMMARY:
The purpose of this voluntary research study is to learn about the potential effects that black raspberry (BRB) lozenges may have on reducing the damage caused from cigarette smoke in mouth cells in adult smokers, which may be useful in reducing health risks associated with smoking.

DETAILED DESCRIPTION:
This clinical trial will consist of a single arm, where participants, after a 1-week baseline period, will be placed on daily BRB administration for a period of 8 weeks followed by a 4 week washout period. Prior to study enrollment, all participants will have an Oral Cancer screening intraoral exam and persons with oral pathology (e.g. premalignant or oral squamous cell carcinoma) will be referred for appropriate clinical care. Biological samples will be collected at 0, 1, 4, 5, 8, 9, 12 and 13 weeks. An 8-week BRB administration period was selected to allow for ample time for effects to be observed in the major endpoints, based on previous clinical data. Likewise, a 4 week washout period at the end of the trial will allow for effects of BRB withdrawal on major outcomes to be measured.

A total of 58 healthy subjects will be recruited into this intervention study. Eligible subjects, after phone screening, will visit the clinic for an additional in-person screening which includes measurement of expired carbon monoxide and pregnancy test (females). Prior to enrollment, each subject will be offered a free oral cancer screening. After obtaining informed consent, eligible subjects will be administered a questionnaire to obtain information on basic demographics, medical history, lifestyle, tobacco and alcohol consumption, and usual dietary intake and biological samples (exfoliated buccal cells and urine) and anthropometric data (e.g. height and weight) will be collected. Subjects will be asked to return after 1 week (Visit 2, 2nd baseline visit) and biological samples will be collected. Subjects will be provided their first supply of test agent (BRB lozenge) and a usage diary and instructed on the proper method for application and completion of the diary entries. At Visits 3-6 (weeks 4, 5, 8, and 9, respectively) subjects will return any unused product, receive a new batch of lozenges (except for week 9), complete a brief questionnaire on compliance and provide biological samples. At week 9 (Visit 6), subjects will return their study diaries and enter the washout period where no test agent will be provided. At the final visits (Visit 7 and 8, weeks 12 and 13), subjects will provide biological samples.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-75
* Smoke 5 cigarettes per day or more for at least the past 12 months
* Have an expired air carbon monoxide measurement of greater than 6 parts per million
* No serious quit attempt in the last one month and not planning to quit in the next 4 months
* Willing and able to attend all study visits
* Able to read and write in English
* Able to understand and provide consent to the study procedures
* Willingness and ability to attend regular visits over a 14-week period and to respond to research contacts between the 5

Exclusion Criteria:

* Unstable or significant medical conditions that affect participant safety or biomarker data in the past 3 months (e.g. recent heart attack, asthma or COPD)
* Women currently pregnant or nursing
* Use of any non-cigarette nicotine delivery product in the past 7 days (e.g. e-cigarettes, pipe or cigar)
* Uncontrolled mental illness or inpatient treatment in the past 6 months; current suicide risk on clinical assessment
* Any known allergy to raspberries
* Use of marijuana or other illegal drugs daily or weekly in the past 3 months
* Use of high dose antioxidant supplements in the past month
* Use of antibiotics
* Heavy drinking (>4 drinks/day, 5 days/week)
* Made no serious cigarette smoking quit attempt or have used any FDA-approved smoking cessation medication in the prior 30 days
* No plan to quit smoking within the next 4 months

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Change of HPB-releasing adducts (buccal cells) from Baseline to end of BRB lozenge treatment at 8 weeks | Baseline, end of 8-week BRB treatment
  Marker of DNA damage caused by tobacco specific nitrosamines in tobacco smoke

SECONDARY OUTCOMES:
Change of B[a]P adducts (buccal cells) from Baseline to end of BRB lozenge treatment at 8 weeks | Baseline, end of 8-week BRB treatment
  Marker of DNA damage caused by benzo[a]pyrene in tobacco smoke
Change of 8-OXO-dG (buccal cells) from Baseline to end of BRB lozenge treatment at 8 weeks | Baseline, end of 8-week BRB treatment
  Biomarker of oxidative damage to DNA caused by tobacco smoke
Change of Anthocyanin (buccal cells) from Baseline to end of BRB lozenge treatment at 8 weeks | Baseline, end of 8-week BRB treatment
  Biomarker of exposure to the black raspberry chemopreventive anthocyanins
Change of Cotinine (urine) from Baseline to end of BRB lozenge treatment at 8 weeks | Baseline, end of 8-week BRB treatment
  Biomarker of tobacco smoke exposure
Change of Creatinine (urine) from Baseline to end of BRB lozenge treatment at 8 weeks | Baseline, end of 8-week BRB treatment
  Biomarker of urine dilution
Change of 8-IsoP (urine) from Baseline to end of BRB lozenge treatment at 8 weeks | Baseline, end of 8-week BRB treatment
  Biomarker of systemic oxidative stress

CONTACTS AND LOCATIONS:
Overall Officials: Karam P El-Bayoumy, Ph.D, Principal Investigator — Penn State University Hershey Medical Center
Locations (1):
- Penn State CTSI Clinical Research Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No